CLINICAL TRIAL: NCT05373693
Title: Evaluation of Visual Performance and Myopia-control Efficacy Afforded by Bestivue Peripheral Defocus Lens (PDL)
Brief Title: Myopia-control Efficacy by Peripheral Defocus Lens (PDL)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TJYYLL-2018-04
Record Dates: First submitted 2022-04-15; First posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-03

CONDITIONS: Myopia, Progressive
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Placebo Comparator): The subjects are randomized to wear SV lens
  Interventions: Device: Single vision lens
- experimental group +2D (Experimental): The subjects are randomized to wear special designed lens with +2D Peripheral Defocus.
  Interventions: Device: +2D PDL
- experimental group +3D (Experimental): The subjects are randomized to wear special designed lens with +3D Peripheral Defocus.
  Interventions: Device: +3D PDL
- experimental group +4D (Experimental): The subjects are randomized to wear special designed lens with +4D Peripheral Defocus.
  Interventions: Device: +4D PDL

INTERVENTIONS:
Device: Single vision lens — Wear single vision lens
  Arms: Control group
Device: +2D PDL — Wear Peripheral defocus lense with +2D
  Arms: experimental group +2D
Device: +3D PDL — Wear Peripheral defocus lense with +3D
  Arms: experimental group +3D
Device: +4D PDL — Wear Peripheral defocus lense with +4D
  Arms: experimental group +4D

SUMMARY:
The proposed study below aims to assess the effect of customized Bestivue PDL lenses on retinal image quality and myopia control. A total of 160 subjected would be enrolled in and randomized to allcoate into four groups. Visual acuity and image blur at various gaze directions and eccentricities on children fitted with +2 to 4 D power and single vision lenses would be measured to assess the short term effect of PDL lens. Axial length and cycloplegic objective refractive error would be measured to assess the Myopia-control Efficacy.

DETAILED DESCRIPTION:
The proposed study below aims to assess the short-term and long-term effect of customized Bestivue PDL lenses on retinal image quality and myopia control. To these ends, two stages of testing are planned. First, objective testing will be utilized to assess the effect of Bestivue PDL lenses on visual acuity and image blur at various gaze directions and eccentricities on 4- to 13-year-old children fitted with +2 to 4 D power and single vision lenses.In the second stage, the same children participants will wear either single or Bestvue PDL lenses with one of the four plus power designs for 2 years. Their corrected visual acuity, objective refractive error with dilation and axial length will be assessed for each eye every six months for two years. Outcomes of these studies should inform whether Bestivue PDL lenses are effective in myopia control while affording adequate visual comfort and performance.

ELIGIBILITY:
Inclusion Criteria:

* The subjects had spherical RE of -1.00 to -6.00 D
* Astigmatism ≤ 4.00 D
* Anisometropia ≤ 1.50 D\
* Best corrected visual acuity (BCVA) equal to or better than logMAR 0.0 (20/20) in both eyes.

Exclusion Criteria:

* Strabismus
* Ocular limitations
* Systemic abnormalities affecting vision and ocular motility.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
changes in cycloplegic objective spherical equivalent (SER) | baseline, 24 months
  changes in cycloplegic objective spherical equivalent (SER) from baseline between four groups.

SECONDARY OUTCOMES:
changes in ocular axial length | baseline, 24 months
  Changes in ocular axial length from baseline between four groups.
visual performance | 1 day
  The visual acuity of peripheral between four groups.

CONTACTS AND LOCATIONS:
Overall Officials: Lihua Li, Principal Investigator — Tianjin Eye Hospital
Locations (1):
- Tianjin Eye Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No